CLINICAL TRIAL: NCT01432691
Title: Clinical and RSA Comparison of Hemi Versus Total Hip Arthroplasty After Displaced Femoral Neck Fracture. A Randomized Double-Blind Study
Brief Title: Hemi Artificial Hipjoint Versus Total Artificial Hipjoint
Acronym: THA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Jakob Klit, MD, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 19761979
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Optimized Treatment
Keywords: Hip-fracture; RSA
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgery (Other): RSA study on hemi
  Interventions: Procedure: Hemi (hemialloplastik)

INTERVENTIONS:
Procedure: Hemi (hemialloplastik) — THA vs hemi
  Other Names: BFX: Biomet CE-number: 00520

SUMMARY:
This is a Randomized Controlled Trial study comparing hemialloplastik versus total joint replacement.

DETAILED DESCRIPTION:
Seventy patients over seventy years who are admitted in our hip fracture department with the indication for hemi joint replacement therapy, due to a Garden 3-4 femoral neck fracture or a fracture Garden 1-2 with over 20-degree posterior tilt are randomized to either hemialloplastik or total joint replacement. The patients are followed for 24 mouths with X-ray Stereo Photogrammetric Analysis (RSA) radiographs and clinical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 70 years, admitted two our hip-fracture department with a 3-4 Garden femoral neck fracture or a fracture Garden 1-2 with over 20-degree posterior tilt.

  * Preoperative New Mobility Score ≥ 6th
* Patients must be able to speak and understand Danish.
* Patients must be able to give informed consent and be cognitively intact (Hindsøe score ≥ 6).
* Patients should be expected to be able to implement the postoperative controls. Patients should not be medically ill: ASA-score ≤ 3rd

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Radiographic and clinical | Five years
  Migration / rotation: Migration is measured by X-ray Stereo Photogrammetric Analysis (RSA).
  Clinical assessment: The patient is assessed clinically using the WOMAC and EQ-5D.

SECONDARY OUTCOMES:
Clinical | Five years
  Implant Placement:
  Mobilisation: Patient mobilization level before the fracture is assessed by the New Mobility Score.Under hospital assessed patients' ability to time with current time instrument daily using the Cumulated ambulation score (CAS).
  Bleeding: Perioperative bleeding set in operation description from start to suture the incision closed. Hgb is measured as standard on the third day in all patients in the hip fracture unit. In addition, registered the need for blood transfusions in the first four postoperative days.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Copenhagen, Copenhagen, Hvidovre, Denmark